CLINICAL TRIAL: NCT03516877
Title: Enhanced Stress Resilience Training for Faculty Physicians
Brief Title: Enhanced Stress Resilience Training for Faculty
Acronym: ESRT-Faculty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-24596
Record Dates: First submitted 2018-04-06; First posted 2018-05-04 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Burnout, Professional
Keywords: Mindfulness-Bases Stress Reduction, Stress, Resilience, Well-being
MeSH Terms: conditions — Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ESRT (Experimental): Volunteer surgery and anesthesia faculty from UCSF working at Parnassus Hospital site and interested in training.
  Volunteer surgery and anesthesia faculty from UCSF working at Zuckerberg San Francisco General Hospital site and interested in training.
  Volunteer surgery and anesthesia faculty from UCSF working at Mission Bay Hospital site and interested in training.
  Interventions: Behavioral: Enhanced Stress Resilience Training for Faculty Physicians

INTERVENTIONS:
Behavioral: Enhanced Stress Resilience Training for Faculty Physicians — Enhanced Stress Resilience Training (ESRT) is derived from Mindfulness-Based Stress Reduction with modifications to language, activities and contextualization to tailor the training to physicians involved in the operating room environment. ESRT consists of 5 weekly 1-hour group classes and 2-4 hour retreat. Classes focus on developing sustained attention and open monitoring in addition to training focused on stress and coping. Increasing duration (3-20 minutes per day) of guided mindfulness exercises are assigned each week. A 2-4 hour intensive retreat occurs at week 4 or 5. The central exercises of the training are the body scan, sitting meditation, qi gong and yoga. The weekly teaching sessions will be offered at various days and times each week in order to accommodate complicated physicians schedules that vary at each site. Participants can attend whichever session is most convenient. Daily practice will occur independently, with the duration reported weekly through text or email.
  Other Names: ESRT

SUMMARY:
Mounting evidence shows that burnout, a critical metric for dissatisfaction and distress, is a growing problem within medicine. Burnout is a syndrome associated with worse physician performance, patient outcomes, and hospital economics. Furthermore, researchers are coming to understand that burnout, diminished performance and the development of mental and physical illness are related. It has been proposed that chronic and overwhelming stress, in the absence of adequate coping skills, promotes performance deficits from surgical errors to poor professionalism due to the effects of stress on cognition.

Notably, in small studies of physicians and other high-stress/high-performance groups mindfulness-based interventions have shown exceptional promise in improving burnout and distress symptoms, protecting cognition, and enhancing meaningfulness and satisfaction in work. Nevertheless, in spite of promising results in various populations the translation of mindfulness-based interventions to real-world settings has been slow.

There is a paucity of quality research examining individually-based interventions, formal mindfulness training in physicians, or either of these things in the high stakes world of surgeons and anesthesiologists. To address these gaps, researchers have developed Enhanced Stress-Resilience Training (ESRT) based on MBSR, but streamlined and tailored for surgeons and anesthesiologists.

Moreover, researchers have refined the scales included in our psychosocial survey of well-being in order to sharpen our approach to the complex issue of physician well-being and factors influencing physician resilience, within Surgery and Anesthesia, at UCSF.

DETAILED DESCRIPTION:
Burnout, which comprises emotional exhaustion, depersonalization and diminished satisfaction with one's work, has been documented in medical students, trainees, and practicing physicians across specialties, including 69% of surgical residents and 40-60% of practicing physicians.

Furthermore, a strong correlation between burnout, impaired performance and the development of mental and physical illness is coming to light. It has been proposed that chronic and overwhelming stress, in the absence of adequate coping skills, promotes burnout and associated distress symptoms such as depression, suicidal ideation and anxiety. Among physicians, performance deficits from surgical errors to poor professionalism have been proposed to result from the effects of stress on cognition. Notably, in other high-stress/high-performance groups, mindfulness-based interventions (MBIs) have shown promise in reducing distress symptoms, protecting cognition, and enhancing performance. Among physicians, limited studies of MBIs have shown improvements in burnout and the sense of meaningfulness and satisfaction in work. Nevertheless, in spite of such evidence, MBIs have yet to be tested in surgeons and have made little progress being translated to real-world settings within healthcare.

Interestingly, our cross-sectional national survey of general surgery residents found that high dispositional mindfulness reduces the risk of emotional exhaustion, depersonalization, moderate to severe depression and suicidal ideation, by 75% or more. This suggests that while mindfulness may seem out of place among surgeons and operating room culture, it is in fact already in use in this setting, albeit unconsciously. More importantly, it appears to be beneficial. These findings, in combination with promising preliminary data from our longitudinal RCT of mindfulness training in surgical interns, suggested that an appropriate MBI could enhance native skills and potentially become a powerful component of stress resilience training among surgeons and anesthesiologists. Therefore, through iterative work in surgical trainees, researchers have created a streamlined, modular MBI for surgery and anesthesia faculty physicians and aim to test it both for pragmatic feasibility and for efficacy at enhancing stress resilience and improving wellbeing.

The significance of this work lies in evaluating a process-centered skill believed to promote resilience, defined as the ability to thrive under adversity and predicated on the perception of stressors as challenges rather than overwhelming threats. The transformation of how people experience stress is a learned skill that can be applied across career stages, practice trajectories and life. The potential to protect individuals, while researchers work for mandatory institutional and systemic change, is powerful. Moreover, the resultant tendency for self-awareness and equipoise has been contagious in other settings, providing fuel for the greater culture change that is inarguably necessary and holds great promise for us and our patients.

The innovation of this work is in bringing a mind-body intervention to bear not only on well-being but also on the fundamental cognitive processes believed to sub-serve performance such as attention, working memory capacity, emotional regulation and self-awareness, which may impact behaviors such as medical decision-making, professionalism and team work. The potential to improve both the operative environment and surgical or medical errors is unprecedented. Moreover, the use of a manualized curriculum specifically crafted for physicians could pave the way for translation to larger studies, other specialties and outside institutions.

ELIGIBILITY:
Exclusion Criteria:

- Lifetime history of an organic mental illness.

Inclusion Criteria:

- Any consented surgery or anesthesia faculty who does not meet exclusion criteria.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Well-being: Burnout | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  Burnout: 2-item Maslach Burnout Inventory, 7-point Likert scale, 0 to 6. High burnout present if either question scores >= 4.
Change in Psychological Well-being: Perceived Stress | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  Cohen's Perceived Stress Scale: 10-items, 5-point Likert scale, 0-4. High stress is score >17.
Change in Psychological Well-being: Anxiety | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  Spielberger's State Trait Anxiety index, 4-point Likert, 1 to 4. High anxiety > 40.
Change in Psychological Well-being: Depression | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  Depression and Suicidal Ideation are assessed using the 9-item form of the Patient Health Questionnaire. 4-point Likert scale, 0 to 3 and a total score from 0 to 27 is calculated. Severe depression > 20.
Change in Psychological Well-being: Mindfulness | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  Cognitive and Affective Mindfulness Scale-Revised. 4-point Likert scale, 1 to 4. High mindfulness ≥ 31.
Change in Psychological Well-being: Alcoholism | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The AUDIT Alcohol Consumption Questions, 5-point Likert scale, 0 to 4. Misuse for females if score ≥ 3, for males if score ≥ 4.
Change in Psychological Well-being: Work Climate | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The Swedish Demand-Control-Support Questionnaire assess work climate. 4-point Likert scale, 1 to 4.
Change in Psychological Well-being: Mental Health | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The short form of the Mental Health Continuum assess various facets of well-being. 6-point Likert scale, 0 to 5.
Change in Psychological Well-being: Perceived Stress Reactivity | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The Perceived Stress Reactivity Scale is a 23-item questionnaire with 5 subscales (Prolonged Reactivity; Reactivity to Work Overload; Reactivity to Social Conflict; Reactivity to Failure; Reactivity to Social Evaluation), and 1 overall scale (Perceived Stress Reactivity total score). The first answer category of each item is coded 0, the second 1, and the third 2.
Change in Psychological Well-being: Mental Disorders | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The Primary Care Evaluation of Mental Disorders Patient Health Questionnaire (PRIME-MD PHQ). This is a 2 item screening instrument used for the assessment of depression with an answer of "yes" to either question indicating a positive response where the respondent displayed traits of possible depression.

SECONDARY OUTCOMES:
Change in Performance: Strategies | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The Test of Performance Strategies-2 is a 68-item self-report instrument that measures a comprehensive range of psychological skills that have been shown to impact successful performance: goal-setting, imagery, self-talk, relaxation, activation, emotional control, and automaticity. 5 point Likert Scale, 1 to 5.
Change in Performance: Psychological Skills | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The Test of Performance Strategies-2 is a 68-item self-report instrument that measures a comprehensive range of psychological skills that have been shown to impact successful performance: goal-setting, imagery, self-talk, relaxation, activation, emotional control, and automaticity. 5 point Likert Scale, 1 to 5.
Change in Emotional Regulation: Mind-Wandering | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The Mind-Wandering Questionnaire, 5 item scale that is measured the frequency of mind-wandering. 6-point Likert scale, 1 to 6. The total is the sum of the five items within a 5-30 range.
Change in Emotional Regulation: Emotions | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The Difficulties in Emotion Regulation Scale, an 18 item scale focuses on adaptive ways of responding to emotional distress. 5-point Likert scale, 1 to 5. The total score is sum the subscale scores.
Change in Emotional Regulation: Decentering | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  The Experiences Questionnaire is a 12 item instrument that assesses decentering. 5-point Likert scale,1 to 5.
Change in Cognitive Function | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  Outcome contains:
  1. NIH EXAMINER Battery. Measures working memory, inhibition, set shifting, fluency, planning, insight, and social cognition and behavior. The EXAMINER battery software calculates the executive composite and factor scores in the R language.
  2. The Cambridge Neuropsychological Test Automated Battery measures:
  1. Reaction Time - assessments of motor and mental response speeds, measures of movement time, reaction time, response accuracy and impulsivity. Outcome measures are divided into reaction time and movement time for both the simple and five-choice variants.
  2. Rapid Visual Information Processing is a measure of sustained attention. Outcome measures cover latency, probability of false alarms and sensitivity.
  3. Paired Associates Learning assesses visual memory and new learning. Outcome measures include the errors made by the participant, the number of trials required to locate the patterns correctly, memory scores and stages completed.
Change in Cognitive Function: NIH EXAMINER Battery | Baseline; 6 weeks (post-intervention); 12 and 18 month follow-up.
  NIH EXAMINER Battery measures working memory, inhibition, set shifting, fluency, planning, insight, and social cognition and behavior. The EXAMINER battery software calculates the executive composite and factor scores in the R language.

CONTACTS AND LOCATIONS:
Overall Officials: Carter C Lebares, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shanafelt TD, Hasan O, Dyrbye LN, Sinsky C, Satele D, Sloan J, West CP. Changes in Burnout and Satisfaction With Work-Life Balance in Physicians and the General US Working Population Between 2011 and 2014. Mayo Clin Proc. 2015 Dec;90(12):1600-13. doi: 10.1016/j.mayocp.2015.08.023. PMID 26653297
- [Result] Shanafelt TD, Balch CM, Bechamps G, Russell T, Dyrbye L, Satele D, Collicott P, Novotny PJ, Sloan J, Freischlag J. Burnout and medical errors among American surgeons. Ann Surg. 2010 Jun;251(6):995-1000. doi: 10.1097/SLA.0b013e3181bfdab3. PMID 19934755
- [Result] Scheepers RA, Boerebach BC, Arah OA, Heineman MJ, Lombarts KM. A Systematic Review of the Impact of Physicians' Occupational Well-Being on the Quality of Patient Care. Int J Behav Med. 2015 Dec;22(6):683-98. doi: 10.1007/s12529-015-9473-3. PMID 25733349
- [Result] Haas JS, Cook EF, Puopolo AL, Burstin HR, Cleary PD, Brennan TA. Is the professional satisfaction of general internists associated with patient satisfaction? J Gen Intern Med. 2000 Feb;15(2):122-8. doi: 10.1046/j.1525-1497.2000.02219.x. PMID 10672116
- [Result] DiMatteo MR, Sherbourne CD, Hays RD, Ordway L, Kravitz RL, McGlynn EA, Kaplan S, Rogers WH. Physicians' characteristics influence patients' adherence to medical treatment: results from the Medical Outcomes Study. Health Psychol. 1993 Mar;12(2):93-102. doi: 10.1037/0278-6133.12.2.93. PMID 8500445
- [Result] Del Canale S, Louis DZ, Maio V, Wang X, Rossi G, Hojat M, Gonnella JS. The relationship between physician empathy and disease complications: an empirical study of primary care physicians and their diabetic patients in Parma, Italy. Acad Med. 2012 Sep;87(9):1243-9. doi: 10.1097/ACM.0b013e3182628fbf. PMID 22836852
- [Result] Sinsky CA, Dyrbye LN, West CP, Satele D, Tutty M, Shanafelt TD. Professional Satisfaction and the Career Plans of US Physicians. Mayo Clin Proc. 2017 Nov;92(11):1625-1635. doi: 10.1016/j.mayocp.2017.08.017. Epub 2017 Nov 1. PMID 29101932
- [Result] Dyrbye LN, Trockel M, Frank E, Olson K, Linzer M, Lemaire J, Swensen S, Shanafelt T, Sinsky CA. Development of a Research Agenda to Identify Evidence-Based Strategies to Improve Physician Wellness and Reduce Burnout. Ann Intern Med. 2017 May 16;166(10):743-744. doi: 10.7326/M16-2956. Epub 2017 Apr 18. No abstract available. PMID 28418518
- [Result] Bodenheimer T, Sinsky C. From triple to quadruple aim: care of the patient requires care of the provider. Ann Fam Med. 2014 Nov-Dec;12(6):573-6. doi: 10.1370/afm.1713. PMID 25384822
- [Result] Campbell J, Prochazka AV, Yamashita T, Gopal R. Predictors of persistent burnout in internal medicine residents: a prospective cohort study. Acad Med. 2010 Oct;85(10):1630-4. doi: 10.1097/ACM.0b013e3181f0c4e7. PMID 20881685
- [Result] Center C, Davis M, Detre T, Ford DE, Hansbrough W, Hendin H, Laszlo J, Litts DA, Mann J, Mansky PA, Michels R, Miles SH, Proujansky R, Reynolds CF 3rd, Silverman MM. Confronting depression and suicide in physicians: a consensus statement. JAMA. 2003 Jun 18;289(23):3161-6. doi: 10.1001/jama.289.23.3161. PMID 12813122
- [Result] Karlamangla AS, Singer BH, McEwen BS, Rowe JW, Seeman TE. Allostatic load as a predictor of functional decline. MacArthur studies of successful aging. J Clin Epidemiol. 2002 Jul;55(7):696-710. doi: 10.1016/s0895-4356(02)00399-2. PMID 12160918
- [Result] Arora S, Sevdalis N, Aggarwal R, Sirimanna P, Darzi A, Kneebone R. Stress impairs psychomotor performance in novice laparoscopic surgeons. Surg Endosc. 2010 Oct;24(10):2588-93. doi: 10.1007/s00464-010-1013-2. Epub 2010 Mar 31. PMID 20354878
- [Result] Wetzel CM, Kneebone RL, Woloshynowych M, Nestel D, Moorthy K, Kidd J, Darzi A. The effects of stress on surgical performance. Am J Surg. 2006 Jan;191(1):5-10. doi: 10.1016/j.amjsurg.2005.08.034. PMID 16399098
- [Result] Jha AP, Stanley EA, Kiyonaga A, Wong L, Gelfand L. Examining the protective effects of mindfulness training on working memory capacity and affective experience. Emotion. 2010 Feb;10(1):54-64. doi: 10.1037/a0018438. PMID 20141302
- [Result] Seppala EM, Nitschke JB, Tudorascu DL, Hayes A, Goldstein MR, Nguyen DT, Perlman D, Davidson RJ. Breathing-based meditation decreases posttraumatic stress disorder symptoms in U.S. military veterans: a randomized controlled longitudinal study. J Trauma Stress. 2014 Aug;27(4):397-405. doi: 10.1002/jts.21936. PMID 25158633
- [Result] Amutio A, Martinez-Taboada C, Delgado LC, Hermosilla D, Mozaz MJ. Acceptability and Effectiveness of a Long-Term Educational Intervention to Reduce Physicians' Stress-Related Conditions. J Contin Educ Health Prof. 2015 Fall;35(4):255-60. doi: 10.1097/CEH.0000000000000002. PMID 26953856
- [Result] Johnson DC, Thom NJ, Stanley EA, Haase L, Simmons AN, Shih PA, Thompson WK, Potterat EG, Minor TR, Paulus MP. Modifying resilience mechanisms in at-risk individuals: a controlled study of mindfulness training in Marines preparing for deployment. Am J Psychiatry. 2014 Aug;171(8):844-53. doi: 10.1176/appi.ajp.2014.13040502. PMID 24832476
- [Result] Lebares CC, Guvva EV, Ascher NL, O'Sullivan PS, Harris HW, Epel ES. Burnout and Stress Among US Surgery Residents: Psychological Distress and Resilience. J Am Coll Surg. 2018 Jan;226(1):80-90. doi: 10.1016/j.jamcollsurg.2017.10.010. Epub 2017 Oct 26. PMID 29107117
- [Result] Wager TD, Davidson ML, Hughes BL, Lindquist MA, Ochsner KN. Prefrontal-subcortical pathways mediating successful emotion regulation. Neuron. 2008 Sep 25;59(6):1037-50. doi: 10.1016/j.neuron.2008.09.006. PMID 18817740
- [Result] Krasner MS, Epstein RM, Beckman H, Suchman AL, Chapman B, Mooney CJ, Quill TE. Association of an educational program in mindful communication with burnout, empathy, and attitudes among primary care physicians. JAMA. 2009 Sep 23;302(12):1284-93. doi: 10.1001/jama.2009.1384. PMID 19773563